CLINICAL TRIAL: NCT01783808
Title: Effects on Exercise Capacity, Physical Activity and Quality of Life Using Ambulatory Oxygen in Patients With Chronic Obstructive Pulmonary Disease (COPD) Who Desaturate Only During Exercise
Brief Title: Intervention Study to Investigate Supplemental Oxygen in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: Umeå University (Other); Karolinska Institutet (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Margareta Emtner, PhD, Associate Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ambox-2012-MEUP; Uppsala University (Other Grant/Funding Number: Uppsala Ethical Review board)
Record Dates: First submitted 2013-01-16; First posted 2013-02-05 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: COPD; Physical Activity; Sedentary
Keywords: COPD; Physical capacity; Physical activity; Inflammatory markers; Health related quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplemental oxygen (Experimental): Patients are supposed to use ambulatory supplemental oxygen during physical activity. The intervention will last for six months.
  In addition to supplemental oxygen the patients will be stimulated by a physiotherapist to be more physically active. A behavioural medicine intervention will be used.
  Interventions: Other: Supplemental oxygen
- Control group (No Intervention): The control group will not get supplemental oxygen during physical activity but they will get the same physical activity intervention as the intervention group.

INTERVENTIONS:
Other: Supplemental oxygen — Patients are supposed to use ambulatory supplemental oxygen during physical activity. The intervention will last for six months.
  In addition to supplemental oxygen the patients will be stimulated by a physiotherapist to be more physically active. A behavioural medicine intervention will be used.
  Arms: Supplemental oxygen

SUMMARY:
The purpose of this trial is to study the effects on exercise capacity, physical activity, inflammatory markers and quality of life of supplemental ambulatory oxygen, to be used during physical activity, in patients with COPD who are normoxic at rest but hypoxemic during a six-min walk test.

Our hypothesis is that if patients are able to use supplemental oxygen they will be more physically active and thereby improve health related quality of life.

DETAILED DESCRIPTION:
Study design The study will employ a parallel design for 6 months including 144 patients (72 patients/group). Patients will be randomized to intervention or control group. The intervention comprises supplemental oxygen to be used during physical activity for 6 months. The control group will receive the same physical activity instructions as the intervention group during the 6 months, but they will not be able to use supplemental oxygen during physical activity.

The study will be a prospective, randomized, single-blind multi-centre intervention study with an intention to treat design (last value carry over). Inclusion will continue until 144 patients have fulfilled the 6 months. Patients will be tested at baseline and after 6 months. There will also be a follow-up after 12 months comprising questionnaires. The study will include centers in Sweden Norway, Finland, and Estonia.

ELIGIBILITY:
Inclusion Criteria:

* COPD, Arterial Oxygen Saturation > 8 kilopascal at rest
* Oxygen Saturation ≤ 88% and a fall in Oxygen Saturation ≥ 4% during a six-minute walk test in ambient air
* No exacerbation within 4 weeks prior to the study
* Post-bronchodilator forced expiratory volume at one second < 80% predicted and forced expiratory volume at one second /Vital capacity < 0.7
* Oxygen Saturation ≥ 92 % during a walk test in self-selected pace with supplemental oxygen. Patients should use supplemental oxygen 10 minutes before the test starts.
* Non-smoker (smoke free for ≥ 6 months)
* Interest in being physically active

Exclusion Criteria:

* Arterial carbon dioxide > 6.5 kilopascal at rest
* Orthopedic, neurologic or mental impairments that would limit physical activity
* Neoplastic disease that is anticipated to influence survival
* Patients exercising with supplemental oxygen
* Long-term oxygen therapy
* Patients with arterial auricular fibrillation and/or heart disease that might hinder physical activity as judged by the physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2012-11 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test | Change from baseline to 6 months
  The patient is supposed to walk as long as possible during six minutes.

SECONDARY OUTCOMES:
Physical activity level | Change from baseline to 6 months
  Physical activity will be measured with an activity monitor (accelerometer) and by a questionnaire

OTHER OUTCOMES:
Health related quality of life | Change from baseline to six months
  EuroQol five-dimension questionnaire, St Georges Respiratory Questionnaire, Hospital Anxiety and Depression Scale, COPD Assessment Test, Medical Research Council scale
Inflammatory markers | Change from baseline to 6 months
  C-reactive protein, Leucocytes, Thrombocytes, Erythrocytes, Hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Christer Janson, Professor, Study Chair — Department of Medical Sciences, Uppsala University
Locations (1):
- Akademiska sjukhuset, Uppsala, Sweden